CLINICAL TRIAL: NCT04494360
Title: Study for the Identification of Participants With Liver Steatosis Who Carry Genetic Variants Associated With Nonalcoholic Fatty Liver Disease (NAFLD)
Brief Title: Study to Estimate How Common it is to Have Genetic Variants Associated With NAFLD
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108830; NOPRODNAS0001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Participants: Healthy participants (men and women) who have, or are likely to have, NAFLD will be enrolled in the study.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No investigational medicinal product will be administered as a part of this study.

SUMMARY:
The purpose of this study is to estimate the prevalence of genetic variants associated with liver disease in participants who are known, or are likely to have NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormality based on medical history, physical exam, and 12-lead electrocardiogram (ECG) collected during Visit 1
* Women must be of non-childbearing potential, defined as either: a.) Postmenopausal or b.) Permanently sterile
* Must be willing to provide a deoxyribonucleic acid (DNA) sample for assessment of genetic variants associated with NAFLD
* Must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study

Exclusion Criteria:

* History or presence of drug abuse within the 2 years prior to Visit 1
* Excessive use of alcohol within 2 years prior to the study
* Body mass index greater than (>) 40 kilogram per meter square (kg/m^2)
* Evidence of other active (acute or chronic) liver disease other than NAFLD/ Nonalcoholic steatohepatitis (NASH)
* History of bariatric surgery or planning to undergo bariatric surgery within the next year
* Inability to undergo magnetic resonance imaging (MRI)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants, who are known to have, or are likely to have, NAFLD.
Sampling Method: Non-Probability Sample
Enrollment: 830 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of Genetic Variants Associated with NAFLD | Up to 8 weeks
  Genotyping for known mutations associated with NAFLD will be conducted and the prevalence in the overall population enrolled will be calculated.
Liver Fat Content Estimated with Fibroscan | Up to 8 weeks
  Fibroscan will be performed to obtain the controlled attenuation parameter (CAP) score to estimate liver fat content. Number of participants with a CAP score greater or equal to (>=) 310 decibels per minute (dB/m) (that is, liver fat >= 10 percent [%]) will be estimated.

SECONDARY OUTCOMES:
Liver Fibrosis Estimated with Fibroscan | Up to 8 weeks
  Fibroscan will be conducted to obtain liver stiffness measurement to estimate liver fibrosis. Number of participants with absent, low or moderate fibrosis (that is, less than or equal to (<=) 9 kilopascals [kPa]) will be estimated.
Hepatic Fat Fraction | Up to 8 weeks
  The liver fat fraction will be obtained by magnetic resonance imaging-proton density fat fraction (MRI-PDFF) to estimate the inter-participant variability in liver fat measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (3):
- United States (3):
  - Research Centers of America, LLC, Hollywood, Florida
  - PRA Health Sciences, Lenexa, Kansas
  - Endeavor Clinical Trials, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency